CLINICAL TRIAL: NCT02775448
Title: Dose-response Study of the Efficacy and Safety of Carduus Marianus in Centesimal Scale for Dyslipidemia in Overweighed or Obese Women in Peri- and Postmenopause: a Randomized Controlled Trial
Brief Title: Dose-response Study of Carduus Marianus in Centesimal Scale for Dyslipidemia in Climacteric Overweighed or Obese Women.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulties in recruiting process
Sponsor: Hospital Nacional Homeopático, Mexico (Other)
Collaborators: Laboratorio Similia, México (Unknown)
Responsible Party: Principal Investigator, Emma del Carmen Macías-Cortés, PhD, Dr., Hospital Nacional Homeopático, Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HospitalNHMexico
Record Dates: First submitted 2016-05-09; First posted 2016-05-17 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Dyslipidemia; Menopause; Obesity
Keywords: Homeopathy; Carduus marianus; Dyslipidemia; Climacteric; Obesity; Triglycerides; Cholesterol; Insulin resistance; LDL-cholesterol; HDL-cholesterol
MeSH Terms: conditions — Dyslipidemias; Obesity; Insulin Resistance | interventions — Exercise; Diet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Diet + exercise + Carduus marianus 6cH (Experimental): Diet (1600 cal/day) + aerobic exercise (30 min daily) + Carduus marianus 6cH, 24 drops diluted in 20 ml of water, by mouth, every 8 hours for 8 weeks.
  Interventions: Drug: Carduus marianus 6cH; Behavioral: Exercise; Other: Diet
- Diet + exercise + Carduus marianus 12cH (Experimental): Diet (1600 cal/day) + aerobic exercise (30 min daily) + Carduus marianus 12cH, 24 drops diluted in 20 ml of water, by mouth, every 8 hours for 8 weeks.
  Interventions: Drug: Carduus marianus 12cH; Behavioral: Exercise; Other: Diet
- Diet + exercise + Carduus marianus 30cH (Experimental): Diet (1600 cal/day) + aerobic exercise (30 min daily) + Carduus marianus 30c, 24 drops diluted in 20 ml of water, by mouth, every 8 hours for 8 weeks.
  Interventions: Drug: Carduus marianus 30cH; Behavioral: Exercise; Other: Diet
- Diet + exercise + placebo (Placebo Comparator): Diet (1600 cal/day) + aerobic exercise (30 min daily) + placebo (87°alcohol), 24 drops diluted in 20 ml of water, by mouth, every 8 hours for 8 weeks.
  Interventions: Drug: Placebo; Behavioral: Exercise; Other: Diet

INTERVENTIONS:
Drug: Carduus marianus 6cH
  Arms: Diet + exercise + Carduus marianus 6cH
Drug: Carduus marianus 12cH
  Arms: Diet + exercise + Carduus marianus 12cH
Drug: Carduus marianus 30cH
  Arms: Diet + exercise + Carduus marianus 30cH
Drug: Placebo
  Arms: Diet + exercise + placebo
Behavioral: Exercise — aerobic exercise, 30 minutes, daily
Other: Diet — 1600 calories

SUMMARY:
Metabolic disorders including hypercholesterolemia and hypertriglyceridemia are present in climacteric women. Carduus marianus is a homeopathic medicine that traditionally has been used for hepatic diseases. It has been used for reducing hypercholesterolemia and hypertriglyceridemia also. The aim of this study is to investigate the most effective dose of Carduus marianus in centesimal scale (6cH, 12cH, 30cH, placebo) plus diet and exercise for reducing hypertriglyceridemia and/or hypercholesterolemia in climacteric women.

DETAILED DESCRIPTION:
The prevalence of metabolic disorders including dyslipidemia increases as women transition from premenopause to postmenopause. This increases the risk for morbidity and mortality from cardiovascular diseases. Carduus marianus is a homeopathic medicine that traditionally has been used for hepatic diseases. Silymarin, isolated from Carduus marianus, owe its therapeutic and hepatoprotective effects to its strong antioxidant and anti-inflammatory properties. Carduus marianus is frequently used in clinical practice and reduces plasma level of triglycerides, total cholesterol and LDL in humans with dyslipidemia. Not all homeopaths agree on dosage and potency when prescribing homeopathic medicines. The aim of this study is to assess: (1) the most effective dose of Carduus marianus in centesimal scale for reducing hypertriglyceridemia and/or hypercholesterolemia in climacteric women; (2) the effect of Carduus marianus in other metabolic parameters (glucose, glycosylated hemoglobin, insulin resistance, weight, body mass index, waist circumference).

This is a 8-week, double-blind, randomized, parallel, four-group, dose-response study to assess the safety and efficacy of Carduus marianus in 6cH, 12cH, 30cH and placebo plus diet and exercise, for reducing hypertriglyceridemia and/or hypercholesterolemia in climacteric women.

ELIGIBILITY:
Inclusion Criteria:

1. women 40-65 years in early or late transition to menopause or postmenopause according to STRAW classification
2. hypertriglyceridemia [>150 <1000 mg/dL], and/or hypercholesterolemia [>200mg/dL]
3. overweight or obesity [BMI >25 Kg/m2]
4. fasting glucose <126mg/dL
5. glycosylated hemoglobin <6.5%
6. be willing and capable to follow study procedures.

Exclusion Criteria:

1. history of cardiovascular disease or coronary risk equivalents
2. secondary hyperlipidemia caused by diabetes mellitus, renal, liver or thyroid diseases
3. hypolipidemic agents, antidiabetic medication, hormone replacement therapy, tamoxifen, raloxifene, danazol, isotretinoin, acitretin, cyclosporin, azathioprine, protease inhibitors (amprenavir, indinavir, nelfinavir, ritonavir, saquinavir), antipsychotics (clozapine), seizure medication (carbamazepine, valproic acid, phenobarbital, phenytoin) either on-going or any time in the previous 2 months
4. any other clinically significant illness that, in the opinion of the investigator, might put the patient at risk of harm during the study or might adversely affect the interpretation of the study data
5. pregnancy or breastfeeding.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline level of triglycerides at 4 and 8 weeks. | 4 and 8 weeks after randomization
Change from baseline level of total cholesterol at 4 and 8 weeks. | 4 and 8 weeks after randomization

SECONDARY OUTCOMES:
Change from baseline level of LDL cholesterol at 4 and 8 weeks. | 4 and 8 weeks after randomization
Change from baseline level of HDL cholesterol at 4 and 8 weeks. | 4 and 8 weeks after randomization
Change from baseline level of fasting glucose at 4 and 8 weeks. | 4 and 8 weeks after randomization
Change from baseline level of glycosylated hemoglobin at 4 and 8 weeks. | 4 and 8 weeks after randomization
Change from baseline [HOMA-IR=insulin(mU/ml) X glucose (mg/dl)/405] at 4 and 8 weeks. | 4 and 8 weeks after randomization
Change from baseline weight (kg) at 4 and 8 weeks. | 4 and 8 weeks after randomization
Change from baseline body mass index (Kg/m2) at 4 and 8 weeks. | 4 and 8 weeks after randomization
Change from baseline waist circumference (cm) at 4 and 8 weeks. | 4 and 8 weeks after randomization
Adverse events | 4 weeks after randomization
  Untoward medical occurrence associated with the use of a drugs in humans, whether or not considered drug related.
Adverse events | 8 weeks after randomization
  Untoward medical occurrence associated with the use of a drugs in humans, whether or not considered drug related.

CONTACTS AND LOCATIONS:
Overall Officials: Emma del Carmen Macias-Cortes, PhD, Principal Investigator — Hospital Nacional Homeopático
Locations (1):
- Hospital Nacional Homeopático, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No